CLINICAL TRIAL: NCT07129161
Title: Iparomlimab and Tuvonralimab Combined With 2 or 4 Cycles of Chemotherapy as Neoadjuvant Therapy for Resectable NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Junye Wang, Chief Physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL-NSCLC-QIBA-1003
Record Dates: First submitted 2025-07-24; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iparomlimab and Tuvonralimab combined with 2 cycles of chemotherapy as neoadjuvant therapy (Experimental): Iparomlimab and Tuvonralimab (5mg/kg Q3W, for 4 cycles) combined with 2 cycles of platinum-based doublet chemotherapy will be administered as neoadjuvant therapy, followed by surgical resection within 6 weeks after completing neoadjuvant therapy. Postoperative adjuvant therapy with the Iparomlimab and Tuvonralimab (5mg/kg, Q3W) for up to 16 cycles may be administered at the investigator's discretion.
  Interventions: Drug: 4 cycles(Iparomlimab and Tuvonralimab 5mg/kg) + 2 cycles (Platinum-based doublet chemotherapy)
- Iparomlimab and Tuvonralimab combined with 4 cycles of chemotherapy as neoadjuvant therapy (Experimental): Iparomlimab and Tuvonralimab (5mg/kg Q3W, for 4 cycles) combined with 4 cycles of platinum-based doublet chemotherapy will be administered as neoadjuvant therapy, followed by surgical resection within 6 weeks after completing neoadjuvant therapy. Postoperative adjuvant therapy with the Iparomlimab and Tuvonralimab (5mg/kg, Q3W) for up to 16 cycles may be administered at the investigator's discretion.
  Interventions: Drug: 4 cycles(Iparomlimab and Tuvonralimab 5mg/kg) + 4 cycles (Platinum-based doublet chemotherapy)

INTERVENTIONS:
Drug: 4 cycles(Iparomlimab and Tuvonralimab 5mg/kg) + 2 cycles (Platinum-based doublet chemotherapy) — Iparomlimab and Tuvonralimab 5mg/kg：5mg/kg，q3W Platinum-based doublet chemotherapy：q3w
  Arms: Iparomlimab and Tuvonralimab combined with 2 cycles of chemotherapy as neoadjuvant therapy
Drug: 4 cycles(Iparomlimab and Tuvonralimab 5mg/kg) + 4 cycles (Platinum-based doublet chemotherapy) — Iparomlimab and Tuvonralimab 5mg/kg：5mg/kg，q3W Platinum-based doublet chemotherapy：q3w
  Arms: Iparomlimab and Tuvonralimab combined with 4 cycles of chemotherapy as neoadjuvant therapy

SUMMARY:
This is a two-arm, randomized, multicenter phase II clinical study to evaluate the efficacy and safety of the Iparomlimab and Tuvonralimab combined with 2 or 4 cycles of chemotherapy as neoadjuvant therapy for resectable stage II-IIIB (N2 only) NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, treatment-naïve Stage II-IIIB (N2 only) non-small cell lung cancer (NSCLC) according to the 9th edition of the American Joint Committee on Cancer (AJCC). Only patients judged as T4 based on tumor size are allowed to be enrolled; other T4 conditions (e.g., invasion of the diaphragm, mediastinal involvement) are not permitted.
* MDT assessment (including a thoracic surgeon) confirms resectability.
* Provision of tumor tissue for biomarker analysis (e.g., PD-L1 testing, gene sequencing).
* At least one measurable lesion per RECIST v1.1.
* ECOG performance status 0 or 1.

Exclusion Criteria:

* Confirmed EGFR or ALK mutations.
* Other malignancies within 5 years (exceptions: adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer post-radical surgery, ductal carcinoma in situ post-radical surgery).
* Prior treatment with immune checkpoint inhibitors (e.g., PD-1/PD-L1 inhibitors, CTLA-4 inhibitors) or immunostimulatory antibodies (e.g., anti-ICOS, CD40, CD137, GITR, OX40), or anti-tumor immune cell therapy.
* Use of immunosuppressants or systemic corticosteroids (>10 mg/day prednisone equivalent) within 2 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | One week postoperatively
  Pathologic complete response (pCR) rate is defined as the percentage of participants with absence of viable tumor cells in the resected lung tumor bed and lymph nodes.

SECONDARY OUTCOMES:
Major Pathologic Response (MPR) Rate | One week postoperatively
  Major pathologic response (MPR) rate is defined as percentage of participants with ≤10% viable tumor cells in the resected lung tumor bed and lymph nodes.
Objective Response Rate (ORR) | Prior to surgery
  Objective Response Rate (ORR) is defined as the percentage of participants with a best response of complete response (CR) or partial response (PR) on preoperative imaging among all subjects who received neoadjuvant therapy and had at least one post-baseline imaging assessment.
R0 Resection rate | At time of surgery
  R0 Resection rate is defined as the percentage of participants who achieve complete surgical resection (R0).
2-Year Event-Free Survival (EFS) Rate | up to 2 years
  EFS is defined as the time from the first study treatment to the occurrence of any event, including disease progression or deterioration preventing surgery, inability to achieve gross resection, disease recurrence, or death from any cause. The 2-year EFS rate was estimated using the Kaplan-Meier method.
Disease-free survival (DFS) | up to 3 years
  Disease-free survival (DFS) is the length of time from postoperative baseline imaging confirmation of no residual disease to disease recurrence or death from any cause, whichever occurs first.
Overall Survival (OS) | up to 3 years
  Overall Survival (OS) is the length of time after initial administration the participant remains alive.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an